CLINICAL TRIAL: NCT02064998
Title: Brief Alcohol Interventions With Mobile Phone Applications for University Students: Interventions Targeting Differing Risk Levels in Two Consecutive Randomized Controlled Trials
Brief Title: Two Consecutive Randomized Controlled Trials Using Mobile Phone Applications for Risky Alcohol Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anne H Berman, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014/278-31/2; KI 2-2439/2014 (PuL) (Other: Karolinska Institutet, Legal Dept.)
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Binge Drinking; Problematic AOD Use
Keywords: Randomized Controlled Trial; Alcohol; Internet; Mobile phone; Screening; Brief intervention
MeSH Terms: conditions — Binge Drinking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Promillekoll (Experimental): Smartphone app monitoring alcohol use with feedback on eBAC level.
  Interventions: Behavioral: Promillekoll
- PartyPlanner (Experimental): Smartphone-adapted web-based app for simulating an event with alcohol consumption in advance, real time monitoring of alcohol use with eBAC feedback during the event and later possibility of comparison between the plan and the event.
  Interventions: Behavioral: PartyPlanner
- Control Study 1 (No Intervention): Waitlist control group that is given access to the Promillekoll and PartyPlanner apps after a 12-week wait.
- Crossover group 1: TeleCoach - Control (Experimental): Six-week access to the TeleCoach app, with exercises and vignettes for reducing or abstaining from alcohol consumption, followed by a 6-week period with no access to the app.
  Interventions: Behavioral: TeleCoach
- Crossover group 2: Control - TeleCoach (Experimental): Initially a 6 week no-app control period, followed by 6-week access to the TeleCoach app, offering exercises and vignettes for reducing or abstaining from alcohol consumption.
  Interventions: Behavioral: TeleCoach

INTERVENTIONS:
Behavioral: Promillekoll — Smartphone app monitoring alcohol use with feedback on eBAC level.
  Arms: Promillekoll
Behavioral: PartyPlanner — Smartphone-adapted web-based app for simulating an event with alcohol consumption in advance, real time monitoring of alcohol use with eBAC feedback during the event and later possibility of comparison between the plan and the event.
  Arms: PartyPlanner
Behavioral: TeleCoach — Smartphone app providing exercises and vignettes for reducing or abstaining from alcohol consumption.
  Arms: Crossover group 1: TeleCoach - Control; Crossover group 2: Control - TeleCoach

SUMMARY:
The purpose of this study is to evaluate the efficacy of three mobile phone applications, Promillekoll, PartyPlanner and TeleCoach among university student union members with problematic drinking. Two trials are conducted, one a three-armed randomized controlled study, and the second a two-armed randomized control study. Outcomes are measured in terms of changes in problematic alcohol use at follow up 6,12 and 18 weeks after baseline data gathering. Both the Promillekoll and PartyPlanner apps feature real time registration of alcohol consumption and give feedback of estimated blood alcohol concentration levels. PartyPlanner also allows for planning an alcohol consumption event in advance and for later comparison of the plan with actual consumption. Study 1 compares these two apps with a control group. In Study 2, participants reporting alcohol consumption above the weekly recommended level are redirected to randomized assignment to an in-depth app, TeleCoach, which offers different exercises for reducing alcohol use. After 6 weeks the controls are offered the TeleCoach intervention for 6 weeks, and the first intervention group loses app access. In both studies, followup occurs 6, 12 and 18 weeks after baseline registration.

Hypotheses:

Study 1: 1. The groups receiving the Promillekoll and PartyPlanner interventions will reduce their alcohol use to a larger extent than the control group at follow-up compared to the baseline level. 2. The planning function in PartyPlanner will be associated with an increased decrease in alcohol consumption compared to only real-time use for Promillekoll.

Study 2: The proportion of participants with risky use above recommended levels will decline faster in the group that receives the intervention first, in comparison to controls.

DETAILED DESCRIPTION:
Objectives:

This is a composite study consisting of Study 1 and Study 2:

Study 1 evaluates the efficacy of two mobile phone applications, Promillekoll and PartyPlanner among university student union members at two or more universities in Sweden. The design is a three-armed randomized controlled trial, and outcomes are measured in terms of changes in problematic alcohol use at followup 6,12 and 18 weeks after baseline data collection. Both Promillekoll and PartyPlanner apps feature real time registration of alcohol consumption and feedback of estimated blood alcohol concentration (eBAC) levels. Both apps show the user when the estimated alcohol level is above 0.6%, a level that can lead to negative health consequences. PartyPlanner additionally provides the possibility of simulating and planning an alcohol consumption event in advance and later on comparing it with consumption at the actual event.

Study 2: At the 6 week followup participants reporting an alcohol consumption above the weekly recommended level in Sweden will be redirected into Study 2. They will be asked to stop using any prior app for alcohol use. Half the group will be randomized to the TeleCoach app intervention, which offers the user different exercises for reducing or abstaining from alcohol use, depending on the user's goal (reduction or abstinence). This group will have access to the app for 6 weeks. The other half of the participants will be randomized to a waitlist control group for 6 weeks. Six weeks into the study, the TeleCoach intervention group will lose access to the app, and the waitlist control group will be given access to the TeleCoach app for 6 weeks.

All participants (in both Study 1 and Study 2) will be followed up at 6, 12 and 18 weeks from initial baseline recruitment.

Method: Study 1:Participants with problematic alcohol use (AUDIT >7 for men and >5 for women), having access to a smartphone running either the Android or the iOs operating systems, are randomized into one of three groups: 1. Access to Promillekoll, 2. Access to PartyPlanner and 3. Waitlist control group (gains access to both apps week 12). Alcohol use outcomes are collected 6,12 and 18 weeks after recruitment to the study.

Study 2: At week 6 of Study 1, participants with risky weekly consumption, i.e. over 9 and 14 Swedish standard glasses (Swedish standard glass = 12 g of alcohol) for women and men respectively are randomized into one of two groups: 1. Access to TeleCoach for 6 weeks, followed by 6 weeks without the app. 2. Six weeks as waitlist controls followed by 6 weeks of access to TeleCoach. Alcohol use outcomes are collected 6 and 12 weeks after entering Study 2 (equivalent to 12 and 18 weeks after initial recruitment to Study 1).

Students without problematic drinking and/or appropriate smartphones also participate in followups, in order to control for the regression to the mean phenomenon. All students who complete all baseline and followup questionnaires participate in a lottery with the chance of winning one of three computer tablets.

Hypotheses:

Study 1: 1. The groups receiving the Promillekoll and PartyPlanner interventions will reduce their alcohol use to a larger extent than the control group at follow-up compared to the baseline level. 2. The planning function in PartyPlanner will be associated with an increased decrease in alcohol consumption compared to only real-time use for Promillekoll.

Study 2: The proportion of participants with risky use above recommended levels will decline faster in the group that receives the intervention first, in comparison to controls.

ELIGIBILITY:
Inclusion Criteria:

* membership in the included student unions

Exclusion Criteria:

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2166 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in estimated Blood Alcohol Concentration (eBAC) | 6, 12 and 18 weeks
  Change in Blood Alcohol Concentration estimated using Widmark's formula for Blood Alcohol Concentration estimation.
Alcohol Use Disorders Identification Test (AUDIT) | 6, 12 and 18 weeks
  Change in total AUDIT score, as a summarized measure of alcohol use (including alcohol consumption and alcohol-related problems).

SECONDARY OUTCOMES:
Quantity | 6, 12 and 18 weeks
  Number of standard drinks consumed over a typical week during last month.
Frequency | 6, 12 and 18 weeks
  Number of drinking occasions over a typical week during the last month

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Berman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska institutet, Department of Clinical Neuroscience, Stockholm, Sweden

REFERENCES:
- [Derived] Gajecki M, Andersson C, Rosendahl I, Sinadinovic K, Fredriksson M, Berman AH. Skills Training via Smartphone App for University Students with Excessive Alcohol Consumption: a Randomized Controlled Trial. Int J Behav Med. 2017 Oct;24(5):778-788. doi: 10.1007/s12529-016-9629-9. PMID 28224445
- [Derived] Berman AH, Gajecki M, Fredriksson M, Sinadinovic K, Andersson C. Mobile Phone Apps for University Students With Hazardous Alcohol Use: Study Protocol for Two Consecutive Randomized Controlled Trials. JMIR Res Protoc. 2015 Dec 22;4(4):e139. doi: 10.2196/resprot.4894. PMID 26693967